CLINICAL TRIAL: NCT00148980
Title: Creation of Bone Marrow Microenvironment for Treatment of MDS in Conjunction With Allogeneic Stem Cell Transplantation
Brief Title: Creation of Bone Marrow Microenvironment for Treatment of Myelodysplastic Syndrome (MDS) in Conjunction With Allogeneic Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 220202-HMO-CTIL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2006-02

CONDITIONS: Myelodysplastic Syndromes; Myelofibrosis
Keywords: Myelodysplastic syndrome (MDS); Allogeneic stem cell transplantation; Demineralized bone matrix (DBM); Bone marrow microenvironment
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis

INTERVENTIONS:
Device: DBM for creation of bone marrow microenvironment

SUMMARY:
Normal bone marrow function depends on the coexistence of normal hematopoietic stem cells and a microenvironment mostly located in the medullary part of the bones. Stem cells cannot function properly in the absence of an adequate microenvironment. Whereas in malignant and non-malignant hematologic diseases caused by a deficiency or abnormal stem cells, stem cell transplantation is the treatment of choice that results in a cure, in diseases such as MDS, myelofibrosis, and other conditions associated with an abnormal microenvironment, pancytopenia may occur despite the presence of apparently normal hematopoietic cells with no recognizable cytogenetic abnormality.

We, the investigators at Hadassah Medical Organization, proved in experimental studies that the entire osteohematopoietic complex consisting of trabecular bone, hematopoietic microenvironment (of stromal origin) and hematopoietic tissue has been successfully transferred directly into ablated bone marrow cavity in a one-step transplantation procedure.

The goal of this study is to enhance hematopoiesis in patients with myelofibrosis syndrome by intraosseous inoculation of demineralized bone matrix (DBM) together with allogeneic bone marrow cells (BMC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with impaired marrow stem cells by cytogenetic analysis or morphology (blasts), considered normal candidates for allogeneic BMT. Such patients will also be entitled to allogeneic bone marrow transplantation with intraosseous DBM.
* Patients with documented myelofibrosis will be entitled to allogeneic bone marrow transplantation with intraosseous DBM.

Exclusion Criteria:

* Patients with anticipated life expectancy of < 4 weeks.
* Pregnant or lactating women.
* Patients with an unrelated disease or relevant clinical problem that may not permit evaluation of the results of the study.
* Patients under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2003-04

PRIMARY OUTCOMES:
Enhancement of hematopoiesis in patients with myelofibrosis MDS by intraosseous demineralized bone matrix together with allogeneic bone marrow transplantation (BMT)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Gurevitch, PhD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel